CLINICAL TRIAL: NCT01783834
Title: Randomized Phase II Study of Pemetrexed Versus Gefitinib in Previously Treated Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Gefitinib Versus Pemetrexed for Previously Treated NSCLC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Eun Kyung Cho, professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-GIRBA-1739
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Previous Treated Metastatic Non-small Cell Lung Cancer
Keywords: Pemetrexed; Gefitinib; iressa; alimta
MeSH Terms: interventions — Gefitinib; Pemetrexed

ARMS (2):
- pemetrexed (Active Comparator): pemetrexed
  Interventions: Drug: Pemetrexed
- gefitinib (Active Comparator): gefitinib
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — compare progression free survivla rate and safety to both drugs
  Other Names: irressa
  Arms: gefitinib
Drug: Pemetrexed — compare PFS rate, safety to both drugs
  Other Names: alimta
  Arms: pemetrexed

SUMMARY:
To compare the efficacy of gefitinib versus pemetrexed as second-line chemotherapy for patients with previous treated non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Cells pathologically diagnosed as histological or radical surgery or radiation therapy is not possible stage IIIB and stage IV non-small-cell lung cancer patients
* second line
* ECOG 0～2
* Patients with normal liver function and renal function

Exclusion Criteria:

* Patients with severe acute infection requiring antibiotic therapy
* Patients who have received treatment in other areas of cancer within 5 years
* During pregnancy and lactation patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 5 years

SECONDARY OUTCOMES:
Progression free survival | 5years

OTHER OUTCOMES:
Number of participants with adverse events | 5years

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon university Gil Medical Center, Incheon, South Korea